CLINICAL TRIAL: NCT04603560
Title: Personalizing Intervention to Reduce Clinical Inertia in the Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nancy Haff, MD, MPH, Associate Epidemiologist, Division of Pharmacoepidemiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020P002897; P30AG064199 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2020-10-27 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This was a cluster-randomized trial randomized at the provider level. Primary care providers were invited to participate and consented into the study. Patients accrued into the study were study-eligible patients cared for by each enrolled primary care provider. The number of participants listed below includes both patients and providers (466 patients and 45 providers).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Audit and Feedback (Experimental): A report of the provider's hypertension control rates compared to benchmark will be displayed using principles of social norming. We will present that provider's hypertension control rates compared to the 90th percentile of their peers.
  Interventions: Behavioral: Audit and Feedback
- Pharmacist E-Detailing (Experimental): A pharmacist will review the chart in advance and provide a personalized recommendation for how to intensify the specific patient's antihypertensive regimen based on current guidelines. For example, they might recommend adding an additional medication based on the patient's comorbid conditions and could suggest a starting dose and timeframe for dose escalation.
  Interventions: Behavioral: Pharmacist E-Detailing
- Control (No Intervention): No intervention will be provided to physicians in the control arm.

INTERVENTIONS:
Behavioral: Audit and Feedback — A report of the provider's hypertension control rates compared to benchmark will be displayed using principles of social norming. We will present that provider's hypertension control rates compared to the 90th percentile of their peers.
  Arms: Audit and Feedback
Behavioral: Pharmacist E-Detailing — A pharmacist will review the chart in advance and provide a personalized recommendation for how to intensify the specific patient's antihypertensive regimen based on current guidelines. For example, they might recommend adding an additional medication based on the patient's comorbid conditions and could suggest a starting dose and timeframe for dose escalation.
  Arms: Pharmacist E-Detailing

SUMMARY:
This is a three-arm pragmatic randomized controlled trial to test two interventions targeting clinical inertia in hypertension compared to control, followed by predictive modeling to identify factors that are associated with intervention responsiveness. Study investigators will use EHR data to identify providers of patients whose hypertension treatment was not intensified. Primary care physicians will then be randomized to one of three arms: pharmacist e-detailing, provider dashboards, or no intervention (control). After the intervention, the investigators will conduct virtual interviews with select providers from each arm. A predictive modeling approach will then be used to identify patient and provider characteristics that are associated with inertia and with responsiveness to each intervention.

DETAILED DESCRIPTION:
We propose a pragmatic randomized controlled trial to test two interventions targeting clinical inertia in hypertension compared to control, followed by predictive modeling to identify factors that are associated with intervention responsiveness.

For Aim 1, we will use Electronic Health Record (EHR) data to identify physicians of patients whose hypertension treatment was not intensified despite their having persistently elevated blood pressure. We will then randomize primary care physicians to on of three arms: academic e-detailing, social norming, or no intervention (control).

For Aim 2, we will conduct interviews with select physicians from each arm. We will then identify patient and physician characteristics that are associated with inertia and with responsiveness to each intervention.

ELIGIBILITY:
Provider Inclusion Criteria:

* Primary care physician
* Practicing in primary care at Massachusetts General Hospital
* Caring for at least 2 patients: (1) aged 18-79, (2) for whom the recent BP history in the last 18 months is above goal, (3) whose most recent BP at an outpatient visit was above goal, and (4) who did not have their hypertension treatment regimens intensified (dose increase, new medication, or medication exchange) at or since that time. The BP goal will be <140/90 for all patients. To accommodate changes in care delivery that occurred during the COVID surge, outpatient visits will include in-office and virtual visits that had vitals recorded in the EHR the same day.

Provider Exclusion Criteria:

* fewer than 100 patients on their primary care panel
* practice less than one session per week

Patient Inclusion Criteria:

* had a blood pressure greater than 140/90 mmHg at 2+ PCP visits in the past 12 months
* treatment was not intensified at any of these visits

Patient Exclusion Criteria:

* excluded from the hypertension registry
* currently pregnant or post-partum 6 months
* receiving hospice care

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haff N, Sreedhara SK, Wood W, Yom-Tov E, Horn DM, Hoover M, Low G, Lauffenburger JC, Chaitoff A, Russo M, Hanken K, Crum KL, Fontanet CP, Choudhry NK. Testing interventions to reduce clinical inertia in the treatment of hypertension: rationale and design of a pragmatic randomized controlled trial. Am Heart J. 2024 Feb;268:18-28. doi: 10.1016/j.ahj.2023.11.005. Epub 2023 Nov 14. PMID 37967641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cluster-randomized trial randomized at the provider level. Primary care providers were invited to participate and consented into the study. Patients accrued into the study were study-eligible patients cared for by each enrolled primary care provider.
Groups:
- Social Norming: Patients: In this arm, patients received care at visits as directed by their primary care providers (PCPs). PCPs received reports that displayed the physician's hypertension control rates compared to their peers.
- Pharmacist E-Detailing: Patients: In this arm, patients received care at visits as directed by their primary care providers (PCPs). PCPs received individual feedback and recommendations generated by a clinical pharmacist delivered as a message through the EHR in advance of eligible patient visits.
- Control: Patients: In this arm, patients received care at visits as directed by their primary care providers (PCPs). No intervention was provided to PCPs in the control arm.
- Social Norming: Providers: In this arm, rates of blood pressure control across all patients with hypertension cared for by each PCP were obtained from a system-wide performance dashboard, and reports were generated that displayed the physician's hypertension control rates compared to their peers. To ensure PCPs were compared to targets that they could reasonably attain, a different comparison was used based on the PCP's current rate of hypertension control. If the PCP's rates were below the practice average, the practice average was used for comparison. If the PCP's rate was above the practice average, the rate of the top performer in the practice was used.
- Pharmacist E-Detailing: Providers: In this arm, PCPs received individual feedback and recommendations generated by a clinical pharmacist delivered as a message through the EHR. Eligible patients with an upcoming (target) visit with their PCP were identified using EHR data, as above. A clinical pharmacist reviewed each patient's chart and generated a personalized recommendation for how to modify the specific patient's antihypertensive regimen based on clinical practice guidelines.
- Control: Providers: No intervention was provided to PCPs in the control arm.
Period: Overall Study
Arm/Group | Social Norming: Patients | Pharmacist E-Detailing: Patients | Control: Patients | Social Norming: Providers | Pharmacist E-Detailing: Providers | Control: Providers
Started (Providers Randomized) | 173 | 143 | 150 | 16 | 15 | 14
Completed (Providers Completed Study) | 173 | 143 | 150 | 16 | 15 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a cluster-randomized trial randomized at the provider level. Primary care providers were invited to participate and consented into the study. Patients accrued into the study were study-eligible patients cared for by each enrolled primary care provider. Baseline demographic characteristics were collected for both patients and providers. Baseline blood pressure was only collected for patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Norming: Patients | Pharmacist E-Detailing: Patients | Control: Patients | Social Norming: Providers | Pharmacist E-Detailing: Providers | Control: Providers | Total
Number analyzed (Participants) | 173 | 143 | 150 | 16 | 15 | 14 | 511
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 64.35 (11.69) | 64.91 (10.72) | 64.11 (12.83) | 53.56 (10.38) | 51.33 (11.1) | 51.71 (13.15) | 64.45 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 75 | 8 | 11 | 10 | 248
  Male | 102 | 70 | 75 | 8 | 4 | 4 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 4 | 20 | 2 | 0 | 0 | 39
  Not Hispanic or Latino | 137 | 129 | 119 | 14 | 15 | 14 | 428
  Unknown or Not Reported | 23 | 10 | 11 | 0 | 0 | 0 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 13 | 10 | 2 | 4 | 4 | 39
  Black or African American | 20 | 17 | 15 | 0 | 1 | 0 | 53
  White | 132 | 105 | 104 | 14 | 9 | 10 | 374
  Other/Unknown/Not reported | 15 | 8 | 21 | 0 | 1 | 0 | 45
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Baseline measurement for patients only. Blood pressures were not obtained for Providers.
  mmHg
    number analyzed (Participants) | 173 | 143 | 150 | 0 | 0 | 0 | 466
    (all) | 148.97 (11.06) | 149.48 (9.02) | 148.13 (10.89) |  |  |  | 148.85 (10.41)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Baseline measurement for patients only. Blood pressures were not obtained for Providers.
  mmHg
    number analyzed (Participants) | 173 | 143 | 150 | 0 | 0 | 0 | 466
    (all) | 81.57 (9.34) | 81.75 (8.82) | 82.78 (8.89) |  |  |  | 82.01 (9.04)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Intensification
Description: The primary outcome was whether physicians intensified treatment at the target visit. Intensification was defined as adding a new antihypertensive medication or increasing the total daily dose of an existing one. This was measured by identifying all prescriptions for anti-hypertensive medications in the electronic health record (EHR) on the day of the target visit and comparing the medication name and total daily dose to anti-hypertensive medications prescribed prior to the target visit date, following the same procedure used to identify intensification during the eligibility assessment
Time Frame: During the primary care office visit in which the provider-patient dyad received the intervention
Measure: Count of Participants; unit: Participants
Groups:
- Social Norming: In this arm, rates of blood pressure control across all patients with hypertension cared for by each PCP were obtained from a system-wide performance dashboard, and reports were generated that displayed the physician's hypertension control rates compared to their peers. To ensure PCPs were compared to targets that they could reasonably attain, a different comparison was used based on the PCP's current rate of hypertension control. If the PCP's rates were below the practice average, the practice average was used for comparison. If the PCP's rate was above the practice average, the rate of the top performer in the practice was used .
- Pharmacist E-Detailing: In this arm, PCPs received individual feedback and recommendations generated by a clinical pharmacist delivered as a message through the EHR. Eligible patients with an upcoming (target) visit with their PCP were identified using EHR data, as above. A clinical pharmacist reviewed each patient's chart and generated a personalized recommendation for how to modify the specific patient's antihypertensive regimen based on clinical practice guidelines.
Arm/Group | Social Norming | Pharmacist E-Detailing | Control
Number analyzed (Participants) | 173 | 143 | 150
Participants | 21 | 23 | 19
Statistical Analysis 1: Comparison: Social Norming vs Control; Generalized estimating equation adjusting for clustering of patients within providers as well as provider panel size; Test type: Superiority; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.54 to 1.66] — The odds ratio represents Social Norming vs Control
Statistical Analysis 2: Comparison: Pharmacist E-Detailing vs Control; Generalized estimating equation adjusting for clustering of patients within providers as well as provider panel size; Test type: Superiority; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.72 to 2.29] — The odds ratio represents Pharmacist E-Detailing vs Control
Statistical Analysis 3: Comparison: Social Norming vs Pharmacist E-Detailing; Generalized estimating equation adjusting for clustering of patients within providers as well as provider panel size; Test type: Superiority; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.74 to 2.56] — The odds ratio represents Pharmacist e-detailing vs Social Norming

ADVERSE EVENTS:
Time Frame: Adverse events were passively collected for patients. Adverse event monitoring began the day each patient entered the study and continued for 9 months.
Description: Because this was a low-risk study conducted within routine primary care, adverse events were monitored passively through information reported to the study team by physician participants as well as through general monitoring of the safety reporting system used within the practices that is reviewed by the study site lead. This monitoring plan was approved by the study's DSMB and reporting was conducted throughout the study.
Groups:
- Social Norming: In this arm, rates of blood pressure control across all patients with hypertension cared for by each PCP were obtained from a system-wide performance dashboard, and reports were generated that displayed the physician's hypertension control rates compared to their peers. To ensure PCPs were compared to targets that they could reasonably attain, a different comparison was used based on the PCP's current rate of hypertension control. If the PCP's rates were below the practice average, the practice average was used for comparison. If the PCP's rate was above the practice average, the rate of the top performer in the practice was used. Adverse events were collected for patients only.
- Pharmacist E-Detailing: In this arm, PCPs received individual feedback and recommendations generated by a clinical pharmacist delivered as a message through the EHR. Eligible patients with an upcoming (target) visit with their PCP were identified using EHR data, as above. A clinical pharmacist reviewed each patient's chart and generated a personalized recommendation for how to modify the specific patient's antihypertensive regimen based on clinical practice guidelines. Adverse events were collected for patients only.
- Control: No intervention will be provided to physicians in the control arm. Adverse events were collected for patients only.
Arm/Group | Social Norming | Pharmacist E-Detailing | Control
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/143 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/143 | 0/150
Other Adverse Events (participants affected / at risk) | 0/173 | 0/143 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04603560/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04603560/ICF_001.pdf